CLINICAL TRIAL: NCT04429685
Title: The Effects of Low Dose Ketamine on Cardiovascular Function
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The focus of the laboratory went a different direction given extramural funding
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Craig Crandall, Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: STU-2019-1792
Record Dates: First submitted 2020-06-04; First posted 2020-06-12 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Healthy
MeSH Terms: interventions — Ketamine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: We plan to implement a crossover design. A parallel design is an alternative approach we may consider as the primary outcome is the effect of low dose ketamine on muscle sympathetic nervous system, for which a placebo administration may not be fully necessary.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low Dose Ketamine (Experimental)
  Interventions: Drug: Ketamine
- Saline (placebo) (Placebo Comparator)
  Interventions: Drug: Saline (placebo)

INTERVENTIONS:
Drug: Ketamine — Low dose ketamine - Ketalar (Racemic Ketamine Hydrochloride) Saline - Isotonic/Normal Saline
  Arms: Low Dose Ketamine
Drug: Saline (placebo) — Saline (placebo)
  Arms: Saline (placebo)

SUMMARY:
Low dose ketamine is used for pain management and for the treatment of anxiety and depression. Prior studies on low dose ketamine have noted short-term (minutes to hours) increases or decreases in blood pressure. Blood pressure that is too high or too low can be problematic if untreated. It is unknown exactly how low dose ketamine affects blood pressure. In fact, no prior studies have measured sympathetic nervous system activity after low dose ketamine has been given to an adult. Because sympathetic nervous system activity has a large influence on blood pressure, we need to know how exactly low dose ketamine affects these body systems. Therefore, in this research we will study how low dose ketamine affects sympathetic nervous system activity and cardiovascular function. The results from this research will inform doctors about how low dose ketamine affects the sympathetic nervous system, heart, and blood vessels.

ELIGIBILITY:
Inclusion Criteria:

* Non-obese (body mass index less than 30 kg/m2)

  *alternatively, individuals will be permitted to participate if they have a body mass index value below 35 kg/m2 but a waist circumference below 88 cm for females and 102 cm for males
* Systolic blood pressure <140 mmHg
* Diastolic blood pressure <90 mmHg

Exclusion Criteria:

* Participants who have cardiac, respiratory, neurological, and/or metabolic illnesses
* Current or previous use of anti-hypertensive medications
* Any known history of renal or hepatic insufficiency/disease
* Pregnancy or breast feeding
* Current smokers, as well as individuals who regularly smoked within the past 3 years
* Individuals with a history of drug abuse
* Individuals who have an unexplained positive urine drug screen (e.g., some agents cause false-positive results, but when the agent is abstained for hours/days/weeks, the repeated drug screen is negative. One example could be an over-the-counter supplement)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2021-05-28 (Actual)

PRIMARY OUTCOMES:
Muscle Sympathetic Nerve Activity Burst Frequency | This outcome will be assessed within one trial lasting up to approximately five hours
  We will measure muscle sympathetic nerve activity (MSNA), quantified as burst frequency and/or incidence, using microneurography

SECONDARY OUTCOMES:
Arterial Blood Pressure | This outcome will be assessed within one trial lasting up to approximately five hours
  We will measure arterial blood pressure, quantified as systolic, mean, and/or diastolic pressure, using an automated monitor before and after administration of low dose ketamine.

OTHER OUTCOMES:
Blood Vessel Diameter | This outcome will be assessed within one trial lasting up to approximately five hours
  We will measure blood vessel function, quantified as blood vessel diameter, using sonography before and after administration of low dose ketamine.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided